CLINICAL TRIAL: NCT02529202
Title: Dexmedetomidine Use During Therapeutic Hypothermia Treatment for Neonates With Hypoxic-ischemic Encephalopathy: The Cool DEX Study
Brief Title: Dexmedetomidine Pharmacokinetics in Neonates During Therapeutic Hypothermia
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Responsible Party: Principal Investigator, Ryan McAdams, Associate Professor of Pediatrics, Neonatologist, Seattle Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15647
Record Dates: First submitted 2015-08-06; First posted 2015-08-20 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2017-01

CONDITIONS: Hypoxic-ischemic Encephalopathy
Keywords: Dexmedetomidine; Neonate; Pharmacokinetics; Therapeutic Hypothermia; Hypoxic-ischemic Encephalopathy; Adrenergic Agents; Adrenergic Agonists; Analgesics; Adrenergic alpha-2 Receptor Agonists; Central Nervous System Agents; Central Nervous System Depressants
MeSH Terms: conditions — Hypoxia-Ischemia, Brain | interventions — Dexmedetomidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dexmedetomidine group (Experimental): Neonates with hypoxic-ischemic encephalopathy will receive a dexmedetomidine maintenance infusion of 0.4 mcg/kg/hr during treatment with therapeutic hypothermia and during re-warming (78 hours total).
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine infusion
  Other Names: Precedex

SUMMARY:
The goal of this proposal is to profile the pharmacokinetics of dexmedetomidine in newborns ≥36 weeks post-menstrual age during therapeutic hypothermia for hypoxic-ischemic encephalopathy.

DETAILED DESCRIPTION:
The goal of this proposal is to determine the pharmacokinetics (PK) of dexmedetomidine (DEX) in newborns in the neonatal intensive care unit (NICU) receiving therapeutic hypothermia (TH) for moderate to severe hypoxic-ischemic encephalopathy (HIE). In newborns with HIE, TH for 72 hours is the standard therapy to mitigate brain damage. Most HIE patients receive mechanical ventilation during TH and are thus sedated with morphine. Unfortunately, morphine has negative side effects and does not specifically prevent shivering. Prevention of shivering is critical to success of TH, as shivering negates cooling. DEX is a particularly promising alternative sedative because it does prevent shivering and is already used in NICUs for sedation and pain management. In newborns, DEX PK data in the setting of TH is not available and needs to be determined to properly dose DEX for HIE patients.

ELIGIBILITY:
Inclusion Criteria:

1. Newborns 36 weeks gestation or older with moderate to severe hypoxic-ischemic encephalopathy identified and treated with therapeutic hypothermia in the Seattle Children's Hospital neonatal intensive care unit.
2. Cooled infants who are initially intubated and mechanically ventilated.
3. Infants anticipated to require 72 hrs of continuous sedation and/or treatment to prevent shivering.
4. Subject's parent(s) or legal guardian(s) has/have voluntarily signed and dated the informed consent document approved by the Institutional Review Board (IRB)/Independent Ethics Committee (IEC).

Exclusion Criteria:

1. Known chromosomal anomalies.
2. Newborns without central lines (e.g., lines not needed or unable to be successfully placed) or without a peripheral arterial line.
3. Patients with known cyanotic congenital heart defects
4. Patients who are participating in another clinical trial.
5. Patients who received DEX prior to enrollment in the study
6. At the discretion of the Investigator, subjects in whom the risk of Dexmedetomidine treatment is expected to exceed its benefits.

Ages: 1 Hour to 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 7 (Actual)
Dates: Start 2016-03; Primary Completion 2016-11 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic (PK) parameter of area under the curve (AUC) | Day 1 to Day 4
  Estimate PK parameter of AUC in newborns ≥36 weeks post-menstrual age with hypoxic-ischemic encephalopathy treated with a continuous dexmedetomidine infusion during therapeutic hypothermia.
Pharmacokinetic (PK) parameter of clearance | Day 1 to Day 4
  Estimate PK parameter of clearance in newborns ≥36 weeks post-menstrual age with hypoxic-ischemic encephalopathy treated with a continuous dexmedetomidine infusion during therapeutic hypothermia.
Pharmacokinetic (PK) parameter of terminal half-life | Day 1 to Day 4
  Estimate PK parameter of terminal half-life in newborns ≥36 weeks post-menstrual age with hypoxic-ischemic encephalopathy treated with a continuous dexmedetomidine infusion during therapeutic hypothermia.
Pharmacokinetic (PK) of volume of distribution | Day 1 to Day 4
  Estimate PK parameter of volume of distribution in newborns ≥36 weeks post-menstrual age with hypoxic-ischemic encephalopathy treated with a continuous dexmedetomidine infusion during therapeutic hypothermia.

SECONDARY OUTCOMES:
Efficacy of dexmedetomidine at preventing shivering | Day 1 to Day 3
  Measure number of morphine doses given for shivering in neonates receiving a continuous dexmedetomidine infusion during therapeutic hypothermia for hypoxic-ischemic encephalopathy.
Safety of dexmedetomidine in neonatal subjects. (composite outcome will include: adverse events, physical examination findings, and vital signs) | Day 1 to Day 4
  Safety assessments will include: adverse events, physical examination findings, vital signs including continuous heart rate, blood pressure, respiratory rate, and pulse oximetry monitoring in neonates receiving a continuous dexmedetomidine infusion during therapeutic hypothermia for hypoxic-ischemic encephalopathy.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan M McAdams, MD, Principal Investigator — Seattle Children's Hospital
Locations (1):
- Seattle Children's Hospital, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No